CLINICAL TRIAL: NCT06447688
Title: The Role of Oral Verapamil in Preventing Radial Spasm During Transradial Angiography
Brief Title: The Role of Verapamil in Radial Artery Spasm
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mersin Medicalpark Hastanesi (Other)
Responsible Party: Principal Investigator, Sefa Sural, MEDICAL DOKTOR( Principal investigator), Mersin Medicalpark Hastanesi
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MLP-SSURAL-001
Record Dates: First submitted 2024-05-31; First posted 2024-06-07 (Actual); Results first posted 2025-10-10 (Actual); Last update posted 2025-10-10 (Actual); Status verified 2025-09

CONDITIONS: Radial Artery Spasm
Keywords: radial artery spasm, verapamil, transradial access
MeSH Terms: interventions — Verapamil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): No other vasodilating drug such as nitrate will be given intravenously
  Interventions: Drug: Verapamil
- Verapamil (Active Comparator): Verapamil will be given orally at least 2 hours before angiography
  Interventions: Drug: Verapamil

INTERVENTIONS:
Drug: Verapamil — Prevent

SUMMARY:
Coronary angiography (CAG) is an invasive imaging method performed to determine the degree of coronary artery disease. Radial artery spasm (RAS) is one of the most common complications during coronary angiography performed via the transradial approach, causing patient discomfort or sometimes interrupting the procedure. There are many studies on RAS, and various pharmacoagents administered intravenously (intraarterial) to prevent RAS have been described. However, there is limited data in the literature regarding oral pharmacoagents that will prevent this complication. In our study, the preventive effect of Verapamil, given orally 2 hours before coronary angiography, on radial artery spasm will be investigated.

DETAILED DESCRIPTION:
Transradial access (TRA) has emerged as the preferred modality for vascular access in coronary interventions worldwide, prompting growing interest in its potential applications across other interventional specialties, especially in neurovascular procedures. Radial artery spasm (RAS) remains the most common complication of TRA, often causing procedural difficulties, patient discomfort, and an increased risk of access site crossover. The incidence of radial artery spasm reported in the literature varies widely, with estimates ranging from 4% to over 51.3%, influenced by factors such as definitions, patient selection, and the operator's experience.

After puncturing the radial artery (Puncture-induced RAS) and inserting the sheath-but before administering intra-arterial spasmolytics-local discomfort and pain may trigger a sympathetic vasoconstrictive response, potentially leading to the onset of RAS.

A previous study has stated that preventing RAS is more effective than treating it after it has been established. In this context, we will conduct a randomized controlled trial to evaluate the efficacy of 120 mg of oral verapamil administered two hours before radial artery puncture in reducing the incidence of radial artery spasm (RAS)

ELIGIBILITY:
Inclusion Criteria:

* Patients who undergo daily coronary angiography
* Whose Allen test is normal.
* Must be able to swallow tablets

Exclusion Criteria:

* Allen test results are distorted,
* No pulse in the radial artery,
* Patients who have previously undergone radial angiography and whose hemodynamics are compromised will be excluded from the study.
* Patients with known contraindications to verapamil (significant aortic stenosis, heart rate <50/min, high-grade atrioventricular block, myocardial infarction) complicated with cardiogenic shock, or left ventricular ejection fraction <35%).

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2024-06-05 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2024-11-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sefa Sural, MD, Principal Investigator — Istinye University
Locations (1):
- VM Medicalpark, Mersin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Sural S, Dogen ME, Duzel B, Karaca O, Brilakis ES, Gorgulu S. The Role of Oral Verapamil in Preventing Radial Spasm During Transradial Angiography. Catheter Cardiovasc Interv. 2025 Aug;106(2):1247-1254. doi: 10.1002/ccd.31675. Epub 2025 Jun 8. PMID 40485154
- See also: Journal publication of study results — https://pubmed.ncbi.nlm.nih.gov/40485154/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All consecutive patients undergoing transradial coronary angiography between June-November 2024 at Medicalpark Hospital (Mersin, Turkey) were included. Exclusion criteria were abnormal Allen test, absent radial pulse, prior radial access, hemodynamic instability, or contraindications to verapamil (e.g., severe AS, HR <50, high-grade AV block, cardiogenic shock, EF <35%).
Pre-assignment Details: No pre-assignment washout or run-in period was required. All eligible participants were randomized immediately after enrollment.
Groups:
- Placebo: Participants did not receive any prophylactic medication to prevent radial artery spasm and underwent standard transradial coronary angiography.
- Verapamil: Participants in this arm received a single oral dose of verapamil (120 mg) prior to the transradial coronary angiography procedure as prophylaxis against radial artery spasm.
Period: Overall Study
Arm/Group | Placebo | Verapamil
Started | 75 | 75
Completed | 75 | 75
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants were included in the analysis
Groups:
- Verapamil: Participants received a single oral dose of verapamil (120 mg) approximately 2 hours before transradial coronary angiography as prophylaxis against radial artery spasm.
- Total: Total of all reporting groups
Arm/Group | Placebo | Verapamil | Total
Number analyzed (Participants) | 75 | 75 | 150
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.1 (12.1) | 59.4 (11.1) | 58.8 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 26 | 49
  Male | 52 | 49 | 101
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Turkey | 75 | 75 | 150

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Clinical Radial Artery Spasm (RAS)
Description: Clinical RAS defined as presence of at least 2 of the following: (1) forearm pain ≥ 4/10, (2) pain during catheter manipulation, (3) catheter movement restriction, (4) pain during sheath removal, (5) difficulty in sheath removal.
Time Frame: During the coronary angiography procedure (up to 2 hours from sheath insertion)
Population: All randomized participants were included in the analysis
Measure: Number; unit: participants
Arm/Group | Placebo | Verapamil
Number analyzed (Participants) | 75 | 75
participants | 23 | 3

2. Primary Outcome: Number of Participants With Ultrasonographically Confirmed Radial Artery Spasm (Ultrasonographic RAS)
Description: Radial artery spasm (RAS) was defined as luminal narrowing of ≥50% as measured by ultrasonography at the access site.
Time Frame: During the procedure, immediately after catheterization (within 2 hours)
Population: All randomized participants were included in the analysis (75 in the placebo group and 75 in the oral verapamil group)
Measure: Number; unit: participants
Groups:
- Placebo: Participants in this group did not receive any prophylactic medication to prevent radial artery spasm
Arm/Group | Placebo | Verapamil
Number analyzed (Participants) | 75 | 75
participants | 36 | 8

3. Secondary Outcome: Number of Participants With Procedural Success
Description: Procedure success was defined as completing coronary angiography or PCI using the initial radial artery approach without requiring a switch to an alternative access site.
Time Frame: During the procedure (from sheath insertion to procedure completion)
Population: All randomized participants were included in the analysis
Measure: Number; unit: participants
Arm/Group | Placebo | Verapamil
Number analyzed (Participants) | 75 | 75
participants | 75 | 75

4. Secondary Outcome: Mean Volume of Contrast Media Used (mL) (mL)
Description: The volume of contrast media (in ml) used was recorded
Time Frame: During the procedure (from sheath insertion to procedure completion)
Population: All randomized participants were included in the analysis
Measure: Mean (Standard Deviation); unit: Milliliters (mL)
Arm/Group | Placebo | Verapamil
Number analyzed (Participants) | 75 | 75
Milliliters (mL) | 133.8 (71.9) | 136.4 (78.3)

5. Secondary Outcome: Mean of the Dose Area Product (DAP)
Description: The parameters collected for radiation exposure included the DAP
Time Frame: During the procedure (from sheath insertion to procedure completion)
Population: All randomized participants were included in the analysis
Measure: Mean (Standard Deviation); unit: Gy·cm2
Arm/Group | Placebo | Verapamil
Number analyzed (Participants) | 75 | 75
Gy·cm2 | 873.9 (732.3) | 878.8 (736.7)

6. Secondary Outcome: Mean of the Fluoroscopy Time
Description: The parameters collected for radiation exposure included the fluoroscopy time (in minutes)
Time Frame: During the procedure (from sheath insertion to procedure completion)
Population: All randomized participants were included in the analysis
Measure: Mean (Standard Deviation); unit: minute
Arm/Group | Placebo | Verapamil
Number analyzed (Participants) | 75 | 75
minute | 7.9 (7.3) | 6.9 (5.8)

ADVERSE EVENTS:
Time Frame: From procedure initiation through hospital discharge (average 1 day)
Description: Adverse events were monitored from the initiation of the coronary angiography procedure through hospital discharge (average 1 day). No deaths, serious adverse events, or non-serious adverse events above the reporting threshold (5%) were observed in either group.
Groups:
- Placebo: Participants in this group did not receive any prophylactic medication to prevent radial artery spasm. They underwent standard transradial coronary angiography without additional vasodilator treatment.
- Verapamil: Participants received a single oral dose of verapamil (120 mg) before the transradial coronary angiography procedure as prophylaxis against radial artery spasm.
Arm/Group | Placebo | Verapamil
All-Cause Mortality (participants affected / at risk) | 0/75 | 0/75
Serious Adverse Events (participants affected / at risk) | 0/75 | 0/75
Other Adverse Events (participants affected / at risk) | 0/75 | 0/75

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-10-24): https://cdn.clinicaltrials.gov/large-docs/88/NCT06447688/Prot_SAP_000.pdf